CLINICAL TRIAL: NCT00580541
Title: Effect of Liking on Fruit Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2023-07
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2007-12

CONDITIONS: Intake of Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: variety — variety and nonvariety

SUMMARY:
Increased dietary variety has been shown to increase intake in animals, as well as humans, as compared to a diet or meal composed of one food. While most studies investigating dietary variety have focused on energy-dense foods (i.e., snack foods) and have emphasized the negative component that variety has on intake, very little research has been conducted with variety to determine if this food characteristic can be used to increase consumption of healthy foods (i.e., fruits). We hypothesize that increasing variety of fruits provided in an eating bout will lead to increased intake of these foods. Therefore, the aim of this investigation is to test the environmental factor of variety on fruit intake in males and females aged 18 to 45 years.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Non-obese
* Unrestrained males and females

Exclusion Criteria:

* Health condition or use medications that influence food intake
* Require specialized diet therapy
* Following a weight loss diet, an athlete, or pregnant or breastfeeding
* Have allergies or aversions to foods used in study
* Report being a binge eater

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
fruit intake | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD, Principal Investigator — University of Tennessee
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States